CLINICAL TRIAL: NCT00519376
Title: A Randomised, Single-dose, Dose Ascending, Double-blind, Placebo Controlled, Four-way, Incomplete Block Crossover Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled Doses of GW642444M With Magnesium Stearate in COPD Patients.
Brief Title: A Study To Investigate The Effect Of Inhaling A Single Dose Of GW642444M In COPD Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2C110165
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2016-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: pharmacodynamics,; Chronic Obstructive Pulmonary Disease (COPD); safety,; COPD patients; pharmacokinetics,; tolerability,; GW642444,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- GW642444M 25mcg (Experimental)
  Interventions: Drug: GW642444M; Drug: placebo
- GW642444M 50mcg (Experimental)
  Interventions: Drug: GW642444M
- GW642444M 100mcg (Experimental)
  Interventions: Drug: GW642444M; Drug: placebo
- GW642444H 100mcg (Experimental)
  Interventions: Drug: GW642444H; Drug: placebo
- placebo (Experimental)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GW642444M — drug
  Arms: GW642444M 100mcg; GW642444M 25mcg; GW642444M 50mcg
Drug: GW642444H — drug
  Arms: GW642444H 100mcg
Drug: placebo
  Arms: GW642444H 100mcg; GW642444M 100mcg; GW642444M 25mcg; placebo

SUMMARY:
This study will involve the use of a new compound, GW642444 that is being developed for the treatment of asthma and chronic obstructive pulmonary disease (COPD). It works by acting on cells in the lungs, causing some of the muscles around the lungs to relax and open up better (bronchodilation), making breathing easier. When a medicine is made into a form ready to be given to patients, the active ingredient is often prepared in the form of a salt, and inactive ingredients (excipients) are often added. Inactive ingredients might be used to help a medicine work better, to make it easier to produce the medicine, or to make it easier to get an accurate dose of medicine. In previous studies the study drug has been given as a dry powder in the form of either the 'H' salt (with the excipient lactose), or in the form of the 'M' salt (with the excipients lactose and cellobiose octaacetate). In this study the 'M' salt form of the study drug has been prepared with lactose and a new excipient called magnesium stearate (instead of cellobiose octaacetate). Participants in this study will receive both the 'H' salt (GW642444H) and the new 'M' salt (GW642444M) containing magnesium stearate. This study will be the first time the new 'M' salt form of the study drug will be given to COPD patients.

ELIGIBILITY:
Inclusion criteria:

* Male or female (of non-childbearing potential) > or = 40 years
* History of COPD
* Smoker or ex-smoker
* Body weight > or = 50 kg with BMI 18-32 kg/m2

Exclusion criteria:

* History of significant disease
* Subjects with a primary asthma diagnosis
* Alpha-1 antitrypsin deficiency as underlying cause of COPD
* Recent respiratory tract infection
* Poorly controlled COPD
* Blood potassium level < 3.5mmol/L
* Short-term or long tern oxygen therapy
* Recent participation in another trial
* History of drug or alcohol abuse
* Known allergies
* Recent blood donation
* ECG abnormalities

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (3):
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kempsford R, Norris V, Siederer S. Vilanterol trifenatate, a novel inhaled long-acting beta2 adrenoceptor agonist, is well tolerated in healthy subjects and demonstrates prolonged bronchodilation in subjects with asthma and COPD. Pulm Pharmacol Ther. 2013 Apr;26(2):256-64. doi: 10.1016/j.pupt.2012.12.001. Epub 2012 Dec 8. PMID 23232038
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: B2C110165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2C110165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C110165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2C110165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2C110165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2C110165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2C110165 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants meeting eligibility criteria at screening were randomized and entered a treatment period. Participants were then randomized to 4 treatment periods in one of 16 sequences (seq) each lasting 1 day and separated by a 7 - 14 day washout period.
Groups:
- Seq 1: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg: Participants were administered single dose of the following treatments: Placebo (PB), GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg. Each participants received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 2: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444M 100 µg: Participants were administered single dose of the following treatments: GW642444M 25 µg, Placebo, GW642444M 50 µg, GW642444M 100 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 3: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444M 100 µg: Participants were administered single dose of the following treatments: GW642444M 25 µg, GW642444M 50 µg, Placebo, GW642444M 100 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 4: GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg, PB: Participants were administered single dose of the following treatments: GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg, Placebo. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 5: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg: Participants were administered single dose of the following treatments: Placebo, GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 6: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444H 100 µg: Participants were administered single dose of the following treatments: GW642444M 25 µg, Placebo, GW642444M 50 µg, GW642444H 100 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 7: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444H 100 µg: Participants were administered single dose of the following treatments: GW642444M 25 µg, GW642444M 50 µg, Placebo, GW642444H 100 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 8: PB, GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg: Participants were administered single dose of the following treatments: Placebo, GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 9: GW642444M 25 µg, PB, GW642444H 100 µg, GW642444M 50 µg: Participants were administered single dose of the following treatments: GW642444M 25 µg, Placebo, GW642444H 100 µg, GW642444M 50 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 10: GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg, PB: Participants were administered single dose of the following treatments: GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg, Placebo. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 11: PB, GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg: Participants were administered single dose of the following treatments: Placebo, GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 12: GW642444M 25 µg, GW642444H 100 µg, PB, GW642444M 50 µg: Participants were administered single dose of the following treatments: GW642444M 25 µg, GW642444H 100 µg, Placebo, GW642444M 50 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 13: GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg, PB: Participants were administered single dose of the following treatments: GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg, Placebo. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 14: GW642444H 100 µg, PB, GW642444M 25 µg, GW642444M 50 µg: Participants were administered single dose of the following treatments: GW642444H 100 µg, Placebo, GW642444M 25 µg, GW642444M 50 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 15: GW642444H 100 µg, GW642444M 25 µg, PB, GW642444M 50 µg: Participants were administered single dose of the following treatments: GW642444H 100 µg, GW642444M 25 µg, Placebo, GW642444M 50 µg. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- Seq 16: GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg, PB: Participants were administered single dose of the following treatments: GW642444H 100 µg, GW642444M 25µg, GW642444M 50 µg, Placebo. Each participant received doses in an ascending dose manner as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
Period: Treatment Period 1
Arm/Group | Seq 1: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg | Seq 2: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444M 100 µg | Seq 3: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444M 100 µg | Seq 4: GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg, PB | Seq 5: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg | Seq 6: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444H 100 µg | Seq 7: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444H 100 µg | Seq 8: PB, GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg | Seq 9: GW642444M 25 µg, PB, GW642444H 100 µg, GW642444M 50 µg | Seq 10: GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg, PB | Seq 11: PB, GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg | Seq 12: GW642444M 25 µg, GW642444H 100 µg, PB, GW642444M 50 µg | Seq 13: GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg, PB | Seq 14: GW642444H 100 µg, PB, GW642444M 25 µg, GW642444M 50 µg | Seq 15: GW642444H 100 µg, GW642444M 25 µg, PB, GW642444M 50 µg | Seq 16: GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg, PB
Started | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Seq 1: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg | Seq 2: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444M 100 µg | Seq 3: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444M 100 µg | Seq 4: GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg, PB | Seq 5: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg | Seq 6: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444H 100 µg | Seq 7: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444H 100 µg | Seq 8: PB, GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg | Seq 9: GW642444M 25 µg, PB, GW642444H 100 µg, GW642444M 50 µg | Seq 10: GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg, PB | Seq 11: PB, GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg | Seq 12: GW642444M 25 µg, GW642444H 100 µg, PB, GW642444M 50 µg | Seq 13: GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg, PB | Seq 14: GW642444H 100 µg, PB, GW642444M 25 µg, GW642444M 50 µg | Seq 15: GW642444H 100 µg, GW642444M 25 µg, PB, GW642444M 50 µg | Seq 16: GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg, PB
Started | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Seq 1: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg | Seq 2: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444M 100 µg | Seq 3: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444M 100 µg | Seq 4: GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg, PB | Seq 5: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg | Seq 6: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444H 100 µg | Seq 7: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444H 100 µg | Seq 8: PB, GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg | Seq 9: GW642444M 25 µg, PB, GW642444H 100 µg, GW642444M 50 µg | Seq 10: GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg, PB | Seq 11: PB, GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg | Seq 12: GW642444M 25 µg, GW642444H 100 µg, PB, GW642444M 50 µg | Seq 13: GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg, PB | Seq 14: GW642444H 100 µg, PB, GW642444M 25 µg, GW642444M 50 µg | Seq 15: GW642444H 100 µg, GW642444M 25 µg, PB, GW642444M 50 µg | Seq 16: GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg, PB
Started | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Unable Evaluate Cardiovascular Endpoints | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Seq 1: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg | Seq 2: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444M 100 µg | Seq 3: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444M 100 µg | Seq 4: GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg, PB | Seq 5: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg | Seq 6: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444H 100 µg | Seq 7: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444H 100 µg | Seq 8: PB, GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg | Seq 9: GW642444M 25 µg, PB, GW642444H 100 µg, GW642444M 50 µg | Seq 10: GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg, PB | Seq 11: PB, GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg | Seq 12: GW642444M 25 µg, GW642444H 100 µg, PB, GW642444M 50 µg | Seq 13: GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg, PB | Seq 14: GW642444H 100 µg, PB, GW642444M 25 µg, GW642444M 50 µg | Seq 15: GW642444H 100 µg, GW642444M 25 µg, PB, GW642444M 50 µg | Seq 16: GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg, PB
Started | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Completed | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Seq 1: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg | Seq 2: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444M 100 µg | Seq 3: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444M 100 µg | Seq 4: GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg, PB | Seq 5: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg | Seq 6: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444H 100 µg | Seq 7: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444H 100 µg | Seq 8: PB, GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg | Seq 9: GW642444M 25 µg, PB, GW642444H 100 µg, GW642444M 50 µg | Seq 10: GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg, PB | Seq 11: PB, GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg | Seq 12: GW642444M 25 µg, GW642444H 100 µg, PB, GW642444M 50 µg | Seq 13: GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg, PB | Seq 14: GW642444H 100 µg, PB, GW642444M 25 µg, GW642444M 50 µg | Seq 15: GW642444H 100 µg, GW642444M 25 µg, PB, GW642444M 50 µg | Seq 16: GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg, PB
Started | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Completed | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Seq 1: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg | Seq 2: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444M 100 µg | Seq 3: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444M 100 µg | Seq 4: GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg, PB | Seq 5: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg | Seq 6: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444H 100 µg | Seq 7: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444H 100 µg | Seq 8: PB, GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg | Seq 9: GW642444M 25 µg, PB, GW642444H 100 µg, GW642444M 50 µg | Seq 10: GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg, PB | Seq 11: PB, GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg | Seq 12: GW642444M 25 µg, GW642444H 100 µg, PB, GW642444M 50 µg | Seq 13: GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg, PB | Seq 14: GW642444H 100 µg, PB, GW642444M 25 µg, GW642444M 50 µg | Seq 15: GW642444H 100 µg, GW642444M 25 µg, PB, GW642444M 50 µg | Seq 16: GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg, PB
Started | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Completed | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Seq 1: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg | Seq 2: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444M 100 µg | Seq 3: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444M 100 µg | Seq 4: GW642444M 25 µg, GW642444M 50 µg, GW642444M 100 µg, PB | Seq 5: PB, GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg | Seq 6: GW642444M 25 µg, PB, GW642444M 50 µg, GW642444H 100 µg | Seq 7: GW642444M 25 µg, GW642444M 50 µg, PB, GW642444H 100 µg | Seq 8: PB, GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg | Seq 9: GW642444M 25 µg, PB, GW642444H 100 µg, GW642444M 50 µg | Seq 10: GW642444M 25 µg, GW642444M 50 µg, GW642444H 100 µg, PB | Seq 11: PB, GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg | Seq 12: GW642444M 25 µg, GW642444H 100 µg, PB, GW642444M 50 µg | Seq 13: GW642444M 25 µg, GW642444H 100 µg, GW642444M 50 µg, PB | Seq 14: GW642444H 100 µg, PB, GW642444M 25 µg, GW642444M 50 µg | Seq 15: GW642444H 100 µg, GW642444M 25 µg, PB, GW642444M 50 µg | Seq 16: GW642444H 100 µg, GW642444M 25 µg, GW642444M 50 µg, PB
Started | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Completed | 2 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GW642444M(25,50 and 100 µg),GW642444H(100 µg), PB in 1-16 Seq: Participants were administered single dose of four of the five following treatments: GW642444M (25, 50 and 100 µg), GW642444H (100 µg) or placebo. Each participant received doses of GW642444M in an ascending dose manner with GW642444H and placebo randomly interspersed as per randomization from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
Arm/Group | GW642444M(25,50 and 100 µg),GW642444H(100 µg), PB in 1-16 Seq
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian/European Heritage | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations. Refer to the General Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the first dose of the study medication until the Follow-up Visit (up to Study Day 60)
Population: All Subjects Population: all participants who received at least one dose of study medication
Measure: Number; unit: Participants
Groups:
- Placebo: Participants received placebo single dose in the morning from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- GW642444M 25 µg: Participants received GW642444M 25 µg single dose in the morning from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- GW642444M 50 µg: Participants received GW642444M 50 µg single dose in the morning from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- GW642444M 100 µg: Participants received GW642444M 100 µg single dose in the morning from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
- GW642444H 100 µg: Participants received GW642444H 100 µg single dose in the morning from the dry powder inhaler (DPI) from the DISKUS/ACCUHALER (one inhalation in the morning).
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 20 | 19 | 8 | 12
Participants
  Any AE | 2 | 1 | 2 | 0 | 0
  Any SAE | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count, and White Blood Cell Count at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count, and white blood cell (WBC) count at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 20 | 19 | 8 | 11
10^9 cells per liter (GI/L)
  Basophils, n=19, 20, 19, 8, 11 | 0.004 (0.0154) | 0.001 (0.0168) | 0.001 (0.0133) | 0.004 (0.0185) | -0.004 (0.0211)
  Eosinophils, n=19, 20, 19, 8, 11 | 0.003 (0.1771) | -0.045 (0.0707) | -0.023 (0.0921) | -0.031 (0.0895) | -0.002 (0.0637)
  Lymphocytes, n=19, 20, 19, 8, 11 | 0.068 (0.4094) | 0.021 (0.3719) | -0.126 (0.2608) | -0.146 (0.4055) | -0.116 (0.3261)
  Monocytes, n=19, 20, 19, 8, 11 | 0.006 (0.1323) | -0.027 (0.1390) | 0.007 (0.0917) | -0.018 (0.1331) | 0.025 (0.1347)
  Total Neutrophils, n=19, 20, 19, 8, 11 | -0.100 (0.6174) | 0.188 (0.9814) | 0.343 (0.9674) | 0.201 (0.6165) | -0.021 (0.7415)
  Platelet count, n=19, 20, 19, 8, 11 | 5.0 (16.16) | 8.2 (18.38) | 8.5 (15.33) | 9.5 (13.72) | -1.1 (10.82)
  WBC, n=19, 20, 19, 8, 11 | -0.02 (0.807) | 0.14 (1.215) | 0.20 (1.029) | 0.04 (1.094) | -0.12 (0.774)

3. Primary Outcome: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of hemoglobin and MCHC at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 20 | 19 | 8 | 11
Grams per liter (g/L)
  Hemoglobin, n=19, 20, 19, 8, 11 | -0.4 (6.21) | -1.2 (6.41) | -0.5 (4.02) | -3.0 (4.21) | 0.8 (5.47)
  MCHC, n=19, 20, 19, 8, 11 | -3.5 (5.23) | -5.8 (22.66) | 1.7 (5.58) | 5.3 (3.65) | -0.8 (6.27)

4. Primary Outcome: Change From Baseline in Reticulocyte and Red Blood Cell (RBC) Count at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of reticulocyte and RBCs at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 20 | 19 | 8 | 11
10^12 cells per liter (TI/L)
  Reticulocytes, n=19, 19, 19, 8, 11 | -0.00714 (0.021416) | -0.00065 (0.019905) | 0.00208 (0.017391) | 0.00905 (0.016387) | 0.00094 (0.012676)
  RBC, n=19, 20, 19, 8, 11 | 0.00 (0.194) | 0.01 (0.193) | -0.01 (0.137) | -0.11 (0.173) | 0.05 (0.186)

5. Primary Outcome: Change From Baseline in Hematocrit at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of hematocrit at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Proportion of 1.0
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 20 | 19 | 8 | 11
Proportion of 1.0 | 0.0044 (0.02025) | -0.0024 (0.02132) | -0.0018 (0.01674) | -0.0161 (0.01408) | 0.0036 (0.02025)

6. Primary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV) at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of MCV at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: Blood samples were collected for the measurement of MCV at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Measure: Mean (Standard Deviation); unit: 10^15 femtoliters (fL) per cell
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 20 | 19 | 8 | 11
10^15 femtoliters (fL) per cell | 0.6 (1.67) | -0.2 (2.09) | -0.2 (1.96) | -1.0 (0.76) | -0.5 (1.81)

7. Primary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) Values at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of MCH at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 picograms (pg) per cell
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 20 | 19 | 8 | 11
10^12 picograms (pg) per cell | -0.11 (0.403) | -0.22 (0.465) | 0.24 (0.581) | 0.14 (0.342) | -0.21 (0.528)

8. Primary Outcome: Change From Baseline in Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Creatine Kinase (CK) and Gamma Glutamyl Transferase (GGT) Values at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of ALT, ALP, AST, and GGT at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: All Subjects Population, Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 17 | 15 | 17 | 7 | 10
International units per liter (IU/L)
  ALT, n=17, 15, 17, 7, 10 | 0.1 (3.89) | -0.5 (2.00) | 1.1 (2.75) | -0.6 (1.51) | 1.0 (4.08)
  ALP, n=17, 15, 17, 7, 10 | 0.4 (10.05) | 1.6 (4.90) | 0.6 (5.93) | -0.4 (2.37) | 1.2 (6.91)
  AST, n=17, 13, 17, 6, 9 | -0.1 (5.46) | -0.6 (2.87) | -1.6 (2.69) | -1.7 (1.03) | 2.1 (5.84)
  GGT, n=17, 15, 17, 7, 10 | -2.0 (2.37) | -0.9 (3.99) | -0.5 (5.06) | -1.6 (2.88) | 0.5 (5.21)
  CK n=17, 15, 17, 7, 10 | -18.1 (29.90) | -20.5 (36.07) | -38.1 (69.67) | -3.1 (15.99) | -19.9 (20.89)

9. Primary Outcome: Change From Baseline in Albumin and Total Protein at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of albumin and total protein at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 17 | 15 | 17 | 7 | 10
Grams per liter
  Albumin, n=17, 15, 17, 7, 10 | -0.9 (2.30) | -0.1 (1.85) | -0.2 (1.51) | -0.9 (1.95) | 0.1 (0.88)
  Total protein, n=17, 15, 17, 7, 10 | -1.7 (4.22) | -0.5 (2.59) | 0.1 (2.34) | -0.7 (3.40) | 0.8 (1.55)

10. Primary Outcome: Change From Baseline in Cholesterol, Chloride, Potassium, Sodium, Triglycerides, and Urea at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of cholesterol, chloride, potassium, sodium, triglycerides, and urea at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 17 | 15 | 17 | 7 | 10
Millimoles per liter (mmol/L)
  Cholesterol, n=17, 15, 17, 7, 10 | -0.085 (0.3416) | 0.121 (0.3764) | 0.032 (1.2588) | -0.251 (0.5630) | 0.082 (0.2447)
  Chloride, n=17, 15, 17, 7, 10 | 0.6 (2.65) | 0.0 (2.80) | -0.3 (2.31) | -0.3 (1.70) | 0.6 (1.43)
  Potassium, n=17, 13, 17, 6, 9 | 0.12 (0.263) | 0.14 (0.384) | 0.06 (0.374) | 0.10 (0.358) | 0.16 (0.305)
  Sodium, n=17, 15, 17, 7, 10 | 0.9 (2.03) | -0.1 (1.83) | 0.4 (1.41) | 0.0 (1.15) | 0.9 (1.79)
  Triglyceride, n=17, 15, 17, 7, 10 | -0.106 (0.4625) | 0.024 (0.5789) | -0.015 (0.3800) | -0.300 (0.5812) | 0.142 (0.2629)
  Urea, n=17, 15, 17, 7, 10 | 0.29 (1.092) | -0.17 (0.964) | -0.38 (1.109) | -0.17 (0.427) | 0.20 (0.918)

11. Primary Outcome: Change From Baseline in Total Bilirubin and Creatinine at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of total bilirubin and creatinine at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 17 | 15 | 17 | 7 | 10
Micromoles per liter (µmol/L)
  Creatinine, n=17, 15, 17, 7, 10 | 3.5 (5.96) | 4.9 (5.62) | 4.9 (6.62) | 1.0 (5.07) | 1.5 (5.28)
  Total Bilirubin, n=17, 15, 17, 7, 10 | -1.1 (2.33) | -0.1 (4.04) | -0.8 (3.60) | 0.3 (1.38) | 1.0 (3.92)

12. Primary Outcome: Change From Baseline in C-reactive Protein at 24 Hours Post-dose on Day 1 of Each Treatment Period
Description: Blood samples were collected for the measurement of c-reactive protein at Baseline and 24 hours post-dose on Day 1of each treatment period. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligrams per liter (Mg/L)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 18 | 18 | 19 | 8 | 10
Milligrams per liter (Mg/L) | -1.36 (3.837) | 0.20 (1.015) | -0.47 (3.500) | -0.76 (2.123) | -0.93 (2.965)

13. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Over the Post-dose 24 Hour (h) Period
Description: SBP and DBP were measured at Baseline and over the post-dose 24 h period at the following scheduled time points: 20 minutes (M), 45 M, 1h, 2h, 3h, 4h, 6h, and 24 h. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 19 | 19 | 8 | 11
Millimeters of mercury (mmHg)
  SBP, 20 M, n=19, 19, 19, 8, 11 | -1.1 (7.20) | -0.6 (6.01) | 1.5 (4.59) | 0.2 (5.38) | -5.2 (8.63)
  SBP, 45 M, n=19, 19, 19, 8, 11 | -1.1 (6.13) | -0.5 (9.16) | -2.6 (8.34) | 1.0 (7.12) | -3.5 (8.23)
  SBP, 1 h, n=19, 19, 19, 8, 11 | -1.0 (8.11) | -0.6 (5.83) | -1.7 (8.46) | -3.1 (10.20) | -4.8 (5.29)
  SBP, 2 h, n=19, 19, 19, 8, 11 | 2.5 (7.77) | -1.2 (9.23) | 0.6 (11.16) | 2.2 (7.73) | -2.7 (6.43)
  SBP, 3 h, n=19, 19, 19, 8, 11 | -0.6 (7.58) | 0.9 (9.75) | 2.6 (7.92) | 4.7 (8.68) | -0.1 (5.60)
  SBP, 4 h, n=19, 19, 19, 8, 11 | 1.1 (6.10) | 0.3 (9.99) | 0.7 (8.18) | 2.2 (7.59) | -0.1 (8.66)
  SBP, 6 h, n=19, 19, 19, 8, 11 | 0.1 (9.41) | -1.4 (10.21) | -0.7 (9.35) | 3.9 (9.82) | -3.2 (9.75)
  SBP, 24 h, n=19, 19, 19, 8, 11 | 0.4 (7.53) | 0.0 (9.01) | -1.8 (8.70) | 3.5 (9.10) | -5.3 (8.21)
  DBP, 20 M, n=19, 19, 19, 8, 11 | -1.9 (4.17) | -0.9 (4.59) | -0.6 (3.95) | 1.3 (1.93) | -4.5 (7.31)
  DBP, 45 M, n=19, 19, 19, 8, 11 | -1.9 (4.65) | -0.1 (6.53) | -3.2 (5.91) | 0.9 (6.63) | -3.8 (5.27)
  DBP, 1 h, n=19, 19, 19, 8, 11 | -2.2 (7.12) | -1.0 (4.46) | -2.3 (4.81) | -0.1 (9.03) | -6.5 (5.99)
  DBP, 2 h, n=19, 19, 19, 8, 11 | 0.2 (6.65) | 0.2 (7.21) | -1.7 (5.73) | 1.3 (6.35) | -3.4 (8.15)
  DBP, 3 h, n=19, 19, 19, 8, 11 | -2.0 (7.32) | -0.0 (5.94) | -1.7 (5.62) | 2.5 (5.10) | -4.0 (7.35)
  DBP, 4 h, n=19, 19, 19, 8, 11 | -2.3 (5.05) | -0.6 (5.15) | -1.7 (5.33) | 1.7 (5.08) | -4.7 (7.76)
  DBP, 6 h, n=19, 19, 19, 8, 11 | -3.2 (7.03) | -0.9 (6.05) | -2.9 (5.05) | -1.1 (5.61) | -7.6 (7.13)
  DBP, 24 h, n=19, 19, 19, 8, 11 | 0.6 (4.49) | -0.5 (5.62) | -1.4 (6.88) | -0.1 (5.38) | -4.1 (6.32)

14. Primary Outcome: Change From Baseline in Heart Rate Over the Post-dose 24 Hour (h) Period
Description: Heart rate (HR) was measured at Baseline and over the post-dose 24 h period at the following scheduled time points: 20 minutes (M), 45 M, 1 h, 2 h, 3 h, 4 h, 6 h, and 24 h. Baseline is defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: Per Protocol (PP) Population: all participants included in the All Subjects population excluding a participant deemed not to have heart rate or other ECG parameters deemed suitable for evaluation. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Beats per minute(bpm)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 19 | 19 | 8 | 11
Beats per minute(bpm)
  20 M, n=19, 19, 19, 8, 11 | -2.9 (4.49) | 0.7 (6.60) | 0.1 (5.58) | 2.2 (6.67) | -2.4 (3.62)
  45 M, n=19, 19, 19, 8, 11 | 0.3 (6.70) | -0.2 (5.51) | 0.3 (5.49) | 4.0 (7.49) | -1.9 (6.70)
  1 h, n=19, 19, 19, 8, 11 | -0.9 (5.33) | -2.1 (5.92) | 0.7 (6.74) | 1.7 (5.36) | -2.2 (5.59)
  2 h, n=19, 19, 19, 8, 11 | 1.6 (7.41) | 3.0 (11.76) | 3.3 (8.34) | 3.0 (7.00) | -0.1 (7.46)
  3 h, n=19, 19, 19, 8, 11 | 1.7 (7.06) | 6.2 (13.76) | 0.7 (8.09) | 2.2 (6.84) | 0.4 (5.43)
  4 h, n=19, 19, 19, 8, 11 | 0.1 (6.57) | 4.8 (13.87) | 2.0 (6.40) | 0.7 (7.72) | 0.1 (6.10)
  6 h, n=19, 19, 19, 8, 11 | 5.7 (10.31) | 2.1 (14.37) | 6.0 (9.32) | 7.4 (11.35) | 3.6 (8.40)
  24 h, n=19, 19, 19, 8, 11 | 1.9 (9.39) | 0.4 (9.05) | 0.2 (6.19) | 0.3 (11.35) | -0.2 (7.91)

15. Primary Outcome: Change From Baseline in Electrocardiographic (ECG) Parameters Over the Post-dose 24 Hour (h) Period
Description: ECG parameters [PR, QRS, RR, QT (uncorrected), QTcB (QT corrected by Bazett's formula) and QTcF (QT corrected by Fridericia's formula) intervals] were measured at Baseline and over the post-dose 24h period at the following scheduled time points: 20 minutes (min), 45 min, 1 h, 2 h, 3 h, 4 h, 6 h, and 24 h. Baseline was defined as the measurement at Screening (Day -28 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: PP Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the PP Population.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 19 | 19 | 8 | 11
milliseconds (msec)
  PR, 20 min, n=19, 19, 19, 8, 11 | -7.3 (17.172) | -1.4 (15.486) | 1.0 (8.650) | 0.5 (11.295) | -8.9 (15.095)
  PR, 45 min, n=19, 19, 19, 8, 10 | -2.7 (7.846) | -3.7 (15.106) | 1.3 (13.588) | -4.5 (12.912) | -4.7 (11.038)
  PR, 1 h, n=19, 19, 19, 8, 11 | -2.8 (17.926) | -2.7 (14.946) | -1.7 (9.511) | 4.3 (19.070) | -3.3 (12.014)
  PR, 2 h, n=19, 19, 19, 8, 11 | -3.3 (12.978) | -1.1 (11.047) | -0.1 (13.800) | -10.1 (44.279) | 2.8 (15.513)
  PR, 3 h, n=19, 19, 19, 8, 11 | 0.1 (12.837) | -3.1 (15.130) | 1.5 (10.602) | 2.8 (20.863) | -3.3 (12.741)
  PR, 4 h, n=19, 19, 19, 8, 11 | -3.0 (13.613) | -1.7 (14.909) | 1.5 (11.102) | 16.98 (25.887) | -2.5 (14.057)
  PR, 6 h, n=18, 19, 19, 8, 11 | -4.0 (10.157) | 0.5 (15.174) | -2.1 (9.437) | 23.59 (21.544) | 3.5 (11.536)
  PR, 24 h, n=19, 19, 18, 8, 11 | -1.4 (18.636) | -1.6 (17.618) | 0.4 (9.101) | 27.07 (20.769) | 2.1 (19.400)
  QRS, 20 min, n=19, 19, 19, 8, 11 | -1.9 (5.031) | -1.0 (3.886) | 0.6 (2.150) | 1.0 (4.719) | 1.4 (4.222)
  QRS, 45 min, n=19, 19, 19, 8, 10 | -1.6 (4.789) | 0.2 (3.928) | 0.2 (3.534) | 0.0 (2.156) | 0.1 (4.601)
  QRS, 1 h, n=19, 19, 19, 8, 11 | -2.0 (5.562) | -0.9 (4.449) | -0.2 (2.155) | 2.7 (4.714) | 1.0 (4.958)
  QRS, 2 h, n=19, 19, 19, 8, 11 | 0.9 (5.393) | -0.3 (3.888) | 0.7 (4.579) | 1.2 (1.265) | -1.0 (6.513)
  QRS, 3 h, n=19, 19, 19, 8, 11 | 0.3 (6.324) | 1.2 (5.194) | 0.3 (3.045) | 0.9 (1.389) | 0.6 (4.670)
  QRS, 4 h, n=19, 19, 19, 8, 11 | -1.0 (4.812) | -0.9 (3.961) | 1.0 (4.937) | 1.0 (4.759) | 1.7 (3.666)
  QRS, 6 h, n=19, 19, 19, 8, 11 | -1.0 (5.156) | -0.1 (4.485) | -0.0 (5.145) | 0.1 (4.254) | 2.0 (4.177)
  QRS, 24 h, n=19, 19, 18, 8, 11 | -1.4 (6.090) | -1.5 (3.736) | 0.7 (2.923) | -0.0 (4.783) | -0.5 (5.546)
  RR, 20 min, n=19, 19, 19, 8, 11 | 48.9 (57.110) | -9.0 (75.077) | 3.9 (73.786) | -29.2 (123.015) | 4.7 (31.266)
  RR, 45 min, n=19, 19, 19, 8, 10 | 5.6 (96.803) | 9.1 (65.366) | -5.7 (81.079) | -73.0 (130.999) | 4.0 (69.539)
  RR, 1 h, n=19, 19, 19, 8, 11 | 29.8 (91.489) | 39.9 (65.636) | -3.7 (84.143) | -29.1 (101.900) | 11.3 (66.621)
  RR, 2 h, n=19, 19, 19, 8, 11 | -0.3 (108.528) | -25.1 (153.206) | -24.2 (127.159) | -29.3 (105.815) | -15.3 (90.415)
  RR, 3 h, n=19, 19, 19, 8, 11 | -12.7 (95.030) | -55.0 (175.742) | 5.6 (129.790) | -35.7 (112.038) | 13.1 (78.368)
  RR, 4 h, n=19, 19, 19, 8, 11 | -21.9 (86.948) | -54.7 (173.646) | -24.6 (85.316) | -17.9 (97.684) | 7.3 (94.243)
  RR, 6 h, n=19, 19, 19, 8, 11 | -61.0 (125.922) | -23.2 (183.705) | -64.1 (127.976) | -106.1 (160.044) | -45.5 (71.133)
  RR, 24 h, n=19, 19, 18, 8, 11 | -4.7 (108.355) | 10.5 (95.865) | 6.0 (103.940) | -1.6 (76.068) | -18.8 (81.880)
  QT, 20 min, n=19, 19, 19, 8, 11 | 4.8 (15.094) | -7.8 (13.891) | -1.7 (9.306) | 2.2 (18.150) | -2.7 (24.051)
  QT, 45 min, n=19, 19, 19, 8, 10 | 5.6 (15.245) | -0.8 (12.037) | -0.1 (11.856) | 2.1 (8.750) | 0.3 (17.997)
  QT, 1 h, n=19, 19, 19, 8, 11 | 5.1 (14.820) | 1.3 (13.453) | 0.5 (13.096) | 2.6 (14.876) | -0.1 (23.941)
  QT, 2 h, n=19, 19, 19, 8, 11 | -4.4 (19.879) | -9.2 (19.465) | -5.6 (18.786) | -10.5 (15.296) | -0.7 (15.403)
  QT, 3 h, n=19, 19, 19, 8, 11 | -5.2 (21.154) | -12.4 (28.408) | 0.8 (18.469) | -10.8 (15.253) | -1.6 (15.403)
  QT, 4 h, n=19, 19, 19, 8, 11 | -7.1 (27.773) | -16.6 (29.661) | -6.3 (14.699) | -5.0 (16.399) | -0.9 (16.693)
  QT, 6 h, n=19, 19, 19, 8, 11 | -17.4 (22.329) | -14.1 (26.540) | -16.9 (20.348) | -20.0 (22.842) | -8.6 (11.990)
  QT, 24 h, n=19, 19, 18, 8, 11 | -9.3 (39.366) | -4.8 (19.461) | 1.1 (30.186) | -0.3 (14.331) | -1.1 (17.099)
  QTc(B), 20 min, n=19, 19, 19, 8, 11 | -5.6 (10.206) | -5.7 (18.465) | -2.5 (13.058) | 7.6 (24.453) | -4.8 (27.410)
  QTc(B), 45 min, n=19, 19, 19, 8, 10 | 4.5 (21.312) | -2.8 (13.737) | 0.9 (13.972) | 18.5 (20.184) | -1.8 (24.471)
  QTc(B), 1 h, n=19, 19, 19, 8, 11 | -0.9 (19.298) | -7.5 (15.779) | 1.2 (12.743) | 7.9 (11.202) | -3.8 (30.201)
  QTc(B), 2 h, n=19, 19, 19, 8, 11 | -4.3 (16.691) | -3.9 (18.963) | 0.0 (16.015) | -4.4 (22.214) | 2.1 (17.456)
  QTc(B), 3 h, n=19, 19, 19, 8, 11 | -1.8 (20.177) | 0.0 (19.550) | 0.4 (20.161) | -3.8 (17.665) | -3.9 (13.908)
  QTc(B), 4 h, n=19, 19, 19, 8, 11 | -0.6 (30.768) | -4.4 (13.490) | -1.3 (11.909) | -1.5 (14.136) | -1.6 (11.578)
  QTc(B), 6 h, n=19, 19, 19, 8, 11 | -3.9 (16.976) | -9.3 (18.612) | -2.9 (15.326) | 3.4 (12.821) | 2.0 (10.667)
  QTc(B), 24 h, n=19, 19, 18, 8, 11 | -9.0 (32.387) | -7.1 (15.386) | -0.2 (14.676) | 0.3 (9.022) | 3.8 (18.294)
  QTc(F), 20 min, n=19, 19, 18, 8, 11 | -2.0 (10.761) | -6.5 (14.867) | -2.2 (9.227) | 5.9 (19.428) | -4.0 (26.022)
  QTc(F), 45 min, n=19, 19, 19, 8, 10 | 4.9 (16.508) | -2.1 (11.430) | 0.6 (9.920) | 13.0 (12.102) | -0.9 (20.795)
  QTc(F), 1 h, n=19, 19, 19, 8, 11 | 1.1 (15.088) | -4.4 (13.387) | 1.0 (9.193) | 6.2 (8.626) | -2.4 (26.900)
  QTc(F), 2 h, n=19, 19, 19, 8, 11 | -4.4 (14.122) | -5.8 (10.606) | -2.0 (11.272) | -6.5 (16.576) | 1.2 (13.750)
  QTc(F), 3 h, n=19, 19, 19, 8, 11 | -3.1 (17.341) | -4.4 (13.383) | 0.5 (14.498) | -6.2 (11.842) | -3.2 (10.836)
  QTc(F), 4 h, n=19, 19, 19, 8, 11 | -3.1 (28.679) | -8.8 (10.344) | -3.0 (9.373) | -2.7 (11.136) | 10.836 (8.648)
  QTc(F), 6 h, n=19, 19, 19, 8, 11 | -8.7 (13.113) | -11.1 (10.871) | -7.8 (10.278) | -4.7 (5.959) | -1.7 (6.561)
  QTc(F), 24 h, n=19, 19, 18, 8, 11 | -9.2 (33.102) | -6.4 (13.364) | 0.0 (17.882) | 0.0 (0.0) | 2.0 (15.496)

16. Secondary Outcome: Mean FEV1 Over 23 and 24 Hours After Dosing
Description: Pulmonary function was measured by forced expiratory volume in one second (FEV1), defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured electronically by spirometry. The data is presented as adjusted mean of the FEV1 values over 23 and 24 hours after dosing. Changed in trough FEV1 will be analysed using a model with baseline, treatment, period, as fixed effects .
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: PP Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Error); unit: Liters
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 17 | 20 | 19 | 6 | 12
Liters | 1.432 (0.0402) | 1.622 (0.0431) | 1.638 (0.0415) | 1.642 (0.0650) | 1.569 (0.0501)

17. Secondary Outcome: Weighted Mean and Maximum Value (0 - 4 Hours) QTc(B) and QTc(F)
Description: QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the 12-lead ECG. QTcB is the QT interval corrected for heart rate using Bazett's formula; QTcF is the QT interval corrected for heart rate using Fridericia's formula. Weighted mean (WM) is derived by calculating the area under curve (AUC), and then dividing by the relevant time interval. QTcB and QTcF recorded at 20 minutes, 45 minutes, 1, 2, 3, and 4 hours post-dose on Day 1 of each treatment period were used for analysis. The data is presented as the adjusted means of WM and maximum QTc(B) and QTc(F).
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: PP Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Error); unit: Milliseconds (msec)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 19 | 19 | 8 | 11
Milliseconds (msec)
  WM QTcB | 419.68 (2.150) | 419.56 (2.378) | 424.18 (2.230) | 422.36 (3.517) | 419.70 (2.714)
  Max QTcB | 439.37 (3.714) | 437.06 (4.104) | 434.62 (3.850) | 438.14 (6.059) | 436.75 (4.681)
  WM QTcF, | 409.13 (1.696) | 408.31 (1.898) | 412.99 (1.760) | 409.50 (2.842) | 409.82 (2.163)
  Max QTcF | 425.34 (2.900) | 421.73 (3.286) | 422.55 (3.025) | 422.41 (5.000) | 422.99 (3.766)

18. Secondary Outcome: Weighted Mean and Maximum Value (0 - 4 Hours) Supine Heart Rate
Description: Weighted mean (WM) is derived by calculating the area under curve (AUC), and then dividing by the relevant time interval. Heart rate was recorded at Screening, prior to dosing, and at 20 minutes, 45 minutes, 1, 2, 3, 4 and 6 hours post-dose on Day 1of each treatment period. Heart rate recorded at 20 minutes, 45 minutes and 1, 2, 3 and 4 hours post-dose on Day 1of the each treatment period were used for analysis. Heart rate measurement was taken in a supine position having rested in this position for at least 10 minutes before each reading. The data is presented as adjusted mean of WM and maximum heart rate.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: PP Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Error); unit: Beats per minute
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 19 | 19 | 8 | 11
Beats per minute
  WM Heart rate | 71.12 (1.320) | 71.76 (1.473) | 71.57 (1.377) | 73.50 (2.179) | 71.22 (1.734)
  Max Heart rate | 77.88 (1.784) | 79.95 (1.948) | 76.13 (1.845) | 77.77 (2.764) | 77.16 (2.248)

19. Secondary Outcome: Weighted Mean and Maximum Value (0 - 4 Hours) of Supine Systolic and Diastolic Blood Pressure
Description: Blood pressure (BP) measurement included systolic blood pressure (SBP) and diastolic BP (DBP). Weighted mean (WM) is derived by calculating the area under curve (AUC), and then dividing by the relevant time interval. SBP and DBP were recorded at Screening, prior to dosing, and at 20 minutes, 45 minutes, 1,2, 3, 4 and 6 hours post-dose on Day 1of the each treatment period. SBP and DBP recorded at 20 minutes, 45 minutes and 1, 2, 3 and 4 hours post-dose on Day 1of the each treatment period were used for analysis. Heart rate measurement was taken in a supine position having rested in this position for at least 10 minutes before each reading. The data is presented as adjusted mean of WM and maximum SBP and DBP.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: PP Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Error); unit: Millimeters of mercury
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 19 | 19 | 19 | 8 | 11
Millimeters of mercury
  WM SBP | 126.92 (1.223) | 126.28 (1.388) | 127.82 (1.284) | 128.99 (2.146) | 125.10 (1.621)
  Max SBP | 133.23 (1.521) | 133.06 (1.714) | 133.91 (1.591) | 135.24 (2.625) | 131.13 (1.994)
  WM DBP | 80.36 (1.017) | 79.74 (1.133) | 80.04 (1.056) | 83.46 (1.721) | 77.46 (1.321)
  Max DBP | 76.13 (1.147) | 75.08 (1.272) | 76.30 (1.189) | 79.92 (1.917) | 71.63 (1.478)

20. Secondary Outcome: Weighted Mean and Maximum/Minimum Value (0 - 4 Hours) for Glucose and Potassium
Description: Blood samples were collected for the measurement of potassium and glucose at Screening, prior to dosing, and at 20 minutes, 45 minutes, 1,2, 3 and 4 hours post-dose on Day 1of the each treatment period. Whole blood samples (approximately 1.0 milliliter [mL]) was analysed for potassium and glucose using the i-STAT1 portable chemical analyser. The i-STAT1 system is an analyser designed for point of care testing and employs a hand-held chemistry analyzer and disposable cartridges, which in the configuration tested, are capable of measuring potassium, glucose, blood gases, electrolytes, metabolites and coagulation. Weighted mean (WM) is derived by calculating the area under curve (AUC), and then dividing by the relevant time interval. The data is presented as adjusted mean of WM and maximum (max) glucose /minimum (min) potassium.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: PP Population. Only those participants available at the indicated time points were assessed.
Measure: Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 17 | 20 | 19 | 6 | 12
Millimoles per liter (mmol/L)
  WM Glucose, n=16,18,19,6,10 | 5.94 (0.204) | 5.86 (0.227) | 5.95 (0.200) | 6.25 (0.345) | 5.71 (0.251)
  Max Glucose, n=17, 20, 19, 6,10 | 6.73 (0.342) | 6.61 (0.370) | 6.65 (0.342) | 6.99 (0.608) | 6.09 (0.436)
  WM Potassium, n=15, 16, 17, 5,12 | 4.29 (0.058) | 4.29 (0.067) | 4.14 (0.057) | 4.22 (0.102) | 4.27 (0.073)
  Min Potassium, n=16, 20, 18, 6,12 | 4.02 (0.052) | 4.03 (0.053) | 3.97 (0.052) | 4.08 (0.082) | 4.08 (0.065)

21. Secondary Outcome: AUC(0- t) and up to 1 Hour Post-dose (AUC[0-1]) of GW642444 and Its Metabolites GI179710, GW630200, and GSK932009, After a Single Dose of GW642444
Description: Blood samples were collected pre-dose and at 2, 5, 10, 20, and 30 minutes, 1, 2, 4, 6, 8, 10, and 24 hour post-dose. Blood samples were analyzed for GW642444 and its metabolites GI179710, GW630200 and GSK932009 using a high performance liquid chromatography/mass spectrometry/mass (HPLC/MS/MS) spectrometry. AUC defined as area under the plasma concentration curve from time zero to the last quantifiable concentration (AUC(0-t)), and up to 1 hour post-dose (AUC(0-1)) were determined by non-compartmental methods. Assay censoring refers to some of the values being below the limit of quantification such that this parameter could not be defined.
Time Frame: Baseline and Day 1 of each treatment period (up to Study Day 54)
Population: Pharmacokinetic (PK) Population: all participants who received at least one dose and for whom a PK sample was obtained and analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms.Hour/milliliter (pg.hr/mL)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 0 | 17 | 19 | 8 | 10
picograms.Hour/milliliter (pg.hr/mL)
  GW642444, AUC(0-t), n=0, 17, 19, 8, 10 |  | 56.49 (86.2) | 222.36 (96.5) | 572.99 (45.3) | 98.13 (0.782)
  GW64244, AUC(0-1), n=0, 11, 18, 8, 10 |  | 58.01 (25.4) | 106.31 (44.5) | 196.24 (23.9) | 54.85 (28.3)
  GI179710, AUC (0-t), n=0, 0, 0, 1, 0 |  | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring.
  GW630200, AUC(0-t), n=0, 0, 0, 0, 0 |  | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring.
  GSK932009, AUC(0-t), n=0, 0, 0, 0, 0 |  | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring.

22. Secondary Outcome: Cmax of GW642444 and Its Metabolites GI179710, GW630200, and GSK932009, After a Single Dose of GW642444
Description: Blood samples were collected pre-dose and at 2, 5, 10, 20, and 30 minutes, 1, 2, 4, 6, 8, 10, and 24 hour post-dose. Blood samples were analyzed for GW642444 and its metabolites GI179710, GW630200 and GSK932009, using a high performance liquid chromatography/mass spectrometry/mass (HPLC/MS/MS) spectrometry. The maximum observed plasma concentration (Cmax) was determined from the concentration time data by non-compartmental methods. Assay censoring refers to some of the values being below the limit of quantification such that this parameter could not be defined.
Time Frame: Day 1 of each treatment period (up to Study Day 54)
Population: PK Population: all participants who received at least one dose and for whom a PK sample was obtained and analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms/milliliter (pg/mL)
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 0 | 20 | 19 | 8 | 12
picograms/milliliter (pg/mL)
  GW642444,n=0, 20, 19, 8, 12 |  | 78.16 (43.9) | 150.60 (53.1) | 259.96 (22.2) | 73.70 (35.7)
  GI179710,n=0, 0, 4, 7, 0 |  | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring.
  GW630200, n=0, 0, 0, 0, 0 |  | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring.
  GSK932009, n=0, 0, 0, 0, 0 |  | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring. | NA (NA) — Insufficient data to define due to assay censoring.

23. Secondary Outcome: Tmax of GW642444 and Its Metabolites GI179710, GW630200, and GSK932009, After a Single Dose of GW642444
Description: Blood samples were collected pre-dose and at 2, 5, 10, 20, and 30 minutes, 1, 2, 4, 6, 8, 10, and 24 hour post-dose. Blood samples were analyzed for GW642444 and its metabolites GI179710, GW630200 and GSK932009, using a high performance liquid chromatography/mass spectrometry/mass (HPLC/MS/MS) spectrometry. The Time to maximum plasma concentration (Tmax) was determined from the concentration time data by non-compartmental methods. Assay censoring refers to some of the values being below the limit of quantification such that this parameter could not be defined.
Time Frame: Day 1 of each treatment period (up to Study Day 54)
Population: PK Population: all participants who received at least one dose and for whom a PK sample was obtained and analyzed
Measure: Median (Full Range); unit: Hours
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Number analyzed (Participants) | 0 | 20 | 19 | 8 | 12
Hours
  GW642444,n=0, 20, 19, 8, 12 |  | 0.175 [0.03 to 2.00] | 0.200 [0.08 to 1.00] | 0.425 [0.15 to 1.03] | 0.500 [0.20 to 2.07]
  GI179710,n=0, 0, 4, 7, 0 |  | NA [NA to NA] — Insufficient data to define due to assay censoring. | 0.140 [0.0 to 0.18] | 0.170 [0.07 to 0.33] | NA [NA to NA] — Insufficient data to define due to assay censoring.
  GW630200, n=0, 0, 0, 0, 0 |  | NA [NA to NA] — Insufficient data to define due to assay censoring. | NA [NA to NA] — Insufficient data to define due to assay censoring. | NA [NA to NA] — Insufficient data to define due to assay censoring. | NA [NA to NA] — Insufficient data to define due to assay censoring.
  GSK932009, n=0, 0, 0, 0, 0 |  | NA [NA to NA] — Insufficient data to define due to assay censoring. | NA [NA to NA] — Insufficient data to define due to assay censoring. | NA [NA to NA] — Insufficient data to define due to assay censoring. | NA [NA to NA] — Insufficient data to define due to assay censoring.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study medication to the end of treatment (up to Study Day 60).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of trial medication during the treatment period.
Arm/Group | Placebo | GW642444M 25 µg | GW642444M 50 µg | GW642444M 100 µg | GW642444H 100 µg
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/19 | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 2/19 | 1/20 | 2/19 | 0/8 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | GW642444M 25 µg (N=20) | GW642444M 50 µg (N=19) | GW642444M 100 µg (N=8) | GW642444H 100 µg (N=12)
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.